CLINICAL TRIAL: NCT05835362
Title: Improving the Outcomes of Adolescents With ADHD Via a Pre-visit Question Prompt List/Video Intervention: a Randomized Controlled Feasibility Trial
Brief Title: Improving the Outcomes of Adolescents With ADHD Via a Pre-visit Question Prompt List/Video Intervention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Health Services Research
Other Study IDs: 22-3288; 1R34MH127139-01A1 (NIH)
Record Dates: First submitted 2023-04-18; First posted 2023-04-28 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: ADHD
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Intervention Model Description: Youth will be randomized within provider to either the question prompt list only group (N=35), the pre-visit video only group (N=35), the combined question prompt list/video intervention group (N=35), or the control group (N=35). This will ensure group balance. The investigators are including a usual care control group because the team needs to control for the many factors that might influence communication (such as youth age, parent educational level, etc.) By randomizing families to the four groups, these factors should be evenly distributed across the groups.
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Question prompt list only group (Experimental): In the question prompt list group youth will be handed the youth ADHD prompt list, and the parent will be handed the parent ADHD prompt list, and will be told, "Your provider wants you to ask any questions that you have about ADHD. Here are lists of questions that you may want to ask. Please spend some time reading through this and marking any questions you want to ask your provider during the visit. You can also write other questions you want to ask on the bottom."
  Interventions: Behavioral: Question prompt list
- Pre-visit video only group (Experimental): Parents and youth in the pre-visit video only group will watch together a short educational video with six themes on an iPad encouraging families to ask questions and to be engaged during ADHD visits.
  Interventions: Behavioral: Pre-visit video
- Combined question prompt list/video intervention group (Experimental): In the combined pre-visit video/question prompt list group youth will watch the video with the parent. Then, youth will be handed the youth ADHD prompt list, and the parent will be handed the parent ADHD prompt list, and will be told, "Your provider wants you to ask any questions that you have about ADHD. Here are lists of questions that you may want to ask. Please spend some time reading through this and marking any questions you want to ask your provider during the visit. You can also write other questions you want to ask on the bottom."
  Interventions: Behavioral: Question prompt list; Behavioral: Pre-visit video; Behavioral: Combined question prompt list/video
- Control group (No Intervention): The control group will receive usual care.

INTERVENTIONS:
Behavioral: Question prompt list — A question prompt list is a list of questions about ADHD (one page) given to study participants to select questions they may want to ask the provider. The youth question prompt list contains 22 questions, and the parent question prompt list contains 20 questions. Both are below a fourth-grade reading level.
  Arms: Combined question prompt list/video intervention group; Question prompt list only group
Behavioral: Pre-visit video — The 11-minute video has six themes: (a) talking to your doctor about ADHD, (b) controlling ADHD without medicine, (c) ADHD medications, (d) ADHD and school, (e) ADHD and your relationships, and (f) helping your parents understand your ADHD.
  Arms: Combined question prompt list/video intervention group; Pre-visit video only group
Behavioral: Combined question prompt list/video — A question prompt list is a list of questions about ADHD (one page) given to study participants to select questions they may want to ask the provider. The youth question prompt list contains 22 questions, and the parent question prompt list contains 20 questions. Both are below a fourth-grade reading level.
  And the video is an 11-minute video that has six themes: (a) talking to your doctor about ADHD, (b) controlling ADHD without medicine, (c) ADHD medications, (d) ADHD and school, (e) ADHD and your relationships, and (f) helping your parents understand your ADHD.
  Arms: Combined question prompt list/video intervention group

SUMMARY:
The investigators propose to conduct a pilot randomized controlled feasibility trial to evaluate the feasibility and effectiveness of a pre-visit intervention to improve communication about attention deficit hyperactivity disorder. The investigators will enroll 140 English-speaking youth ages 11-17 with an ADHD medical record diagnosis who screen as having predominantly inattentive subtype, hyperactive/impulsive subtype, or combined inattention/hyperactivity on the Vanderbilt parent assessment scale from three pediatric clinics. Teh investigators will randomize the families to receive both the question prompt lists and video (N=35), just the question prompt lists (N=35), just the video (N=35), or usual care (N=35). This will allow the team to understand whether both the video and question prompt list components are needed for the larger trial. The aims of the investigators are:

Aim 1: To examine whether the ADHD question prompt lists and/or pre-visit video significantly impact the proposed mechanisms of the intervention. The team will investigate whether adolescents and parents in each of the intervention groups: (a) ask more questions and receive more provider education about ADHD during their baseline and 3-month visits and (b) have higher self-efficacy at 3 and 6 months than adolescents and parents in the usual care group.

Aim 2: To investigate the effectiveness of the ADHD question prompt lists and/or the pre-visit video by examining whether adolescents in each of the intervention groups have improved ADHD symptoms, school and social performance, and quality-of-life at 6 months compared to those in the usual care group.

Aim 3: To assess adolescent, parent, and provider feedback on the acceptability, feasibility, tolerability, and safety of using the ADHD question prompt lists and/or the pre-visit video. The results from this pilot trial will be used to inform a larger trial by: (a) identifying the intervention arm with the greatest potential impact, acceptability, feasibility, and tolerability, and (b) determine the best mechanisms and outcome variables to assess in a larger trial.

DETAILED DESCRIPTION:
Using Social Cognitive Theory as a guide, the investigators hypothesize that an ADHD video/question prompt list intervention will increase youth and parent question-asking which, in turn, will increase provider education during the medical visit, which ultimately will improve youth and parent ADHD self-efficacy. Youth and parent question asking, provider education, and self-efficacy are the proposed mechanisms of the intervention. By improving youth and parent self-efficacy to manage ADHD, the investigators also hypothesize that youth ADHD symptoms, school and social performance, and quality-of-life will improve.

The investigators propose to conduct a pilot randomized controlled feasibility trial to evaluate the feasibility and effectiveness of a pre-visit intervention to improve communication about ADHD. The team will enroll 140 English-speaking youth ages 11-17 with an ADHD medical record diagnosis who screen as having predominantly inattentive subtype, hyperactive/impulsive subtype, or combined inattention/hyperactivity on the Vanderbilt parent assessment scale from three pediatric clinics. The investigators will randomize the families to receive both the question prompt lists and video (N=35), just the question prompt lists (N=35), just the video (N=35), or usual care (N=35). This will allow us to understand whether both the video and question prompt list components are needed for the larger trial. The aims of the investigators are:

Aim 1: To examine whether the ADHD question prompt lists and/or pre-visit video significantly impact the proposed mechanisms of the intervention. The team will investigate whether adolescents and parents in each of the intervention groups: (a) ask more questions and receive more provider education about ADHD during their baseline and 3 month visits and (b) have higher self-efficacy at 3 and 6 months than adolescents and parents in the usual care group.

Aim 2: To investigate the effectiveness of the ADHD question prompt lists and/or the pre-visit video by examining whether adolescents in each of the intervention groups have improved ADHD symptoms, school and social performance, and quality-of-life at 6 months compared to those in the usual care group.

Aim 3: To assess adolescent, parent, and provider feedback on the acceptability, feasibility, tolerability, and safety of using the ADHD question prompt lists and/or the pre-visit video. The results from this pilot trial will be used to inform a larger trial by: (a) identifying the intervention arm with the greatest potential impact, acceptability, feasibility, and tolerability, and (b) determine the best mechanisms and outcome variables to assess in a larger trial.

The investigators will conduct this study at three pediatric clinics. The principal investigator will enroll 30 providers from three participating pediatric clinics. Those providers who are interested will complete a consent form and a short demographic questionnaire. Eligible patients of participating providers will be called by clinic staff who will explain the study. The clinic staff will ask interested families to arrive 20 minutes before their next visit to meet with a research assistant to learn more about the study. The investigators will enroll 140 youth (approximately 40 to 60 from each clinic). The UNC research staff will explain the study. The research assistant will take the family to a private area within the clinic to learn more about the study. The research assistant will obtain parent informed consent, parent permission, and youth assent. Parents will be asked to complete HIPAA forms. Then the research assistant will administer the eligibility screener. Youth will be randomized to either the question prompt list only group (N=35), the pre-visit video only group (N=35), the combined question prompt list/video intervention group (N=35), or the control group (N=35), stratified by provider. This will ensure group balance. Using a random number generator, the biostatistician will prepare opaque, sealed envelopes containing group assignments. The research assistant will open the envelope when a youth enrolls into the study. Youth and parents in question prompt list group will be handed the prompt lists and will be told, "Your provider wants you to ask any questions that you have about ADHD. Here are lists of questions that you may want to ask. Please spend some time reading through this and marking any questions you want to ask your provider during the visit. You can also write other questions you want to ask on the bottom." Parents and youth in the pre-visit video only group will watch a short educational video with six themes on an iPad encouraging families to ask questions and to be engaged during ADHD visits. Youth and parents in the combined pre-visit video/question prompt list group will watch the video and will then be handed the question prompt lists and given the instructions above. The control group will receive usual care.

Next, all participating families (both the intervention and control group families) will have their medical visits audio-tape recorded. After the medical visit, the research assistant will conduct a 15- to 20-minute interview with all participating youth while parents complete a questionnaire. For those in the question prompt list or combined video/question prompt list intervention groups, the research assistant will collect the youth's and parent's question prompt lists so that the investigators can compare what questions the youth and parent wanted to ask to what the youth and parent asked during the visit.

Youth typically come back for ADHD follow-up visits every 3 months. Families in the intervention groups will receive the intervention to which the families were randomly assigned to use at each follow-up visit. The research assistant will interview all youth and have the parent complete a questionnaire after the 3- and 6-month visits. The research assistant will audiotape the 3 month visit since the investigators will be examining how baseline and 3-month communication is associated with 6-month outcomes. The youth's medical records will be reviewed for ADHD diagnosis date, co-morbidities, number of ADHD visits, and ADHD treatment use (medications and other strategies) for the 6-month period before enrollment into the study and the 6-month period after.

Youth will receive a small stipend for each interview and parents will receive a small stipend as well for completing the questionnaire at each time point (baseline, 3 months, and 6 months). The investigators will ask teachers to complete the Vanderbilt symptoms and performance assessments at baseline, 3 months, and 6 months. Teachers will receive a small stipend at each data collection point.

Towards the end of the trial, the investigators will hold a lunchtime meeting with the providers at each clinic and ask the teachers to complete validated and reliable measures of intervention acceptability, feasibility, and tolerability for each intervention group (question prompt lists, video, question prompt lists and video). The providers will each receive a small stipend for their time. The adolescents in the intervention groups will complete the acceptability, feasibility, and tolerability questions at the 6-month interviews and the parents will complete them in the 6-month questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Youth eligibility criteria are: age 11 to 17 years, speak and read English, have an ADHD diagnosis, are present for an ADHD visit, and screen as having predominantly inattentive subtype, hyperactive/impulsive subtype, or combined inattention/hyperactivity on the Vanderbilt parent assessment scale. Youth's parents will be eligible if they are at least 18 years of age, speak and read English, and are the legal guardian of the child.

Exclusion Criteria:

* Child does not have ADHD.
* Child is not between the ages of 11 and 17.
* Child does not see a provider at the clinic who is participating in the study.
* Child does not speak English.
* Child/parent does not want to have today's medical visit audio-recorded.
* Parent under 18 years of age, do not speak and read English, and are not the legal guardian of the adolescent.

Ages: 11 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 126 (Actual)
Dates: Start 2023-03-22 (Actual); Primary Completion 2025-11-30 (Actual); Study Completion 2025-11-30 (Actual)

PRIMARY OUTCOMES:
Vanderbilt Assessment Total Symptom Score (parent informant) | 6 months
  The Vanderbilt parent informant ADHD rating scales is a Diagnostic and Statistical Manual for Mental Disorders-IV-based scale, which give a Total Symptom Score. The Vanderbilt ADHD Rating Scale has been shown to have valid psychometric properties consistent with the Diagnostic and Statistical Manual for Mental Disorders; the Vanderbilt includes all the DSM-IV symptoms for ADHD. The Vanderbilt has demonstrated acceptable internal consistency, adequate factor structure, and good reliability and validity as a measure of youth behavior and school functioning. The Vanderbilt includes 18 DSM-IV symptoms that are rated on a 4-point Likert scale ranging from 0 to 3. The parent (primary outcome) Total Symptom Scores (TSS) will be calculated by summing the scores on each item; summary scores can range from 0 to 54. Higher scores indicate worse symptoms. The investigators will examine changes in the total symptom summary score from baseline to 6 months.
Youth functioning using the Vanderbilt Assessment (parent informant) Average Performance Score | 6 months
  The Vanderbilt average performance score (parent informant) has 8 functional impairment items (overall school performance, reading, writing, math, relationship with parents, relationship with siblings, relationship with peers, and participation in organized activities such as team sports) measured on a 5-point Likert scale (ranging from 1 to 5). A summary score will be calculated by summing the scores and dividing by the 8 items to calculate an average performance score. Higher scores indicate worse performance. The investigators will examine changes in the average performance score from baseline to 6 months.

CONTACTS AND LOCATIONS:
Overall Officials: Betsy Sleath, PhD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- University of North Carolina at Chapel Hill, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual data that supports the final trial results will be shared beginning 9 to 36 months following publication provided the investigator who proposes to use the data has approval from an Institutional Review Board (IRB), Independent Ethics Committee (IEC), or Research Ethics Board (REB), as applicable, and executes a data use/sharing agreement with UNC. Because this is a vulnerable population only specific de-identified data that preserves confidentiality to the extent allowed by NIMH will be shared.
Time Frame: Beginning 9 and continuing for 36 months following publication
Access Criteria: Investigator has approved IRB, IEC, or REB and an executed data use/sharing agreement with UNC.

DOCUMENTS (1):
  • Informed Consent Form (2022-12-20): https://cdn.clinicaltrials.gov/large-docs/62/NCT05835362/ICF_000.pdf